CLINICAL TRIAL: NCT01881022
Title: An Evaluation of an Internet-based, Psychosexual Intervention for Couples Following Treatment for Breast Cancer: A Phase I Trial
Brief Title: An Internet-based Psychosexual Intervention for Couples Following Treatment for Breast Cancer
Acronym: IPSIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Canadian Breast Cancer Foundation (Other)
Responsible Party: Principal Investigator, Karen Fergus, Principal Investigator, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CBCF-092013
Record Dates: First submitted 2013-06-14; First posted 2013-06-19 (Estimated); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Couples; Sexual Dysfunction; Psychosexual Intervention; Sex Therapy; Online Support; e-health
MeSH Terms: conditions — Breast Neoplasms; Sexual Dysfunction, Physiological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Psychosexual Intervention (Experimental): The intervention will consist of 6 weekly sessions of couples psychosexual counseling delivered via videoconferencing.
  Interventions: Behavioral: Psychosexual Intervention

INTERVENTIONS:
Behavioral: Psychosexual Intervention — Couples will complete six weekly psychosexual counselling sessions. Each session will focus on areas relevant to sex therapy and sexual dysfunction in couples facing breast cancer (e.g. education, communication, body imagery, sensate focusing, and problem solving). Sessions will be one hour in length (Note: Session 1 will be 1.5 hours), during which couples will meet with a facilitator via videoconferencing.

SUMMARY:
Diagnosis and treatment of breast cancer often leads to lower levels of sexual desire, decreased sexual arousal, painful intercourse, and difficulties achieving orgasm, and thus adversely impacts sexual functioning and intimacy. Despite the overwhelming evidence that many couples experience sexual distress following breast cancer, very few interventions have been designed exclusively to address these concerns. The purpose of this study is to develop and evaluate an online psychosexual program geared to the unique needs of couples experiencing sexual distress after breast cancer. This study will utilize a web-based approach, allowing couples to participate in the program from the privacy and comfort of their homes, and providing a resource to couples who may not otherwise be able to readily access support. Accordingly, this project has the potential for widespread positive impact for couples affected by breast cancer.

DETAILED DESCRIPTION:
Many couples experience sexual problems following breast cancer treatment, and difficulties with intimacy and sexuality tend to extend past the 1 year post-treatment point. Given that resources available for couples who experience sexual distress after breast cancer are virtually non-existent, there is a need to develop and empirically evaluate psychosexual interventions for breast cancer patients and their partners.

The purpose of this study is to evaluate the feasibility, process, and outcomes of an online, couples-based intervention designed to address sexual problems encountered by many couples facing breast cancer. The intervention will take place in the form of six E-therapy sessions delivered via secure, encrypted videoconferencing software commonly used by health care providers practicing telemedicine. Each session will be supplemented by psychoeducational materials (i.e. reading and/or video) available through a privately accessed homepage for the study.

Thirty couples will participate in the study, and will be be randomized to either the treatment condition or the wait-list control condition. Participants assigned to the wait-list will have the option of receiving the online program once they have completed their commitment to the study (approximately 5 months later). In addition to completing standardized questionnaires, couples will participate in pre- and post-treatment interviews, which will be analyzed thematically in order to improve the intervention and its delivery.

The proposed project builds upon existing research pertaining to the sexual health implications of female cancer survivorship, and will fill a gap both in the literature and support available to breast cancer survivors experiencing sexual distress. Given that sexual distress is such a crucial concern for women with breast cancer, and that the majority of couples experiencing sexual difficulties may not receive adequate support in this regard, the goal of the proposed project will be the creation of an accessible, cost-effective, empirically validated tool that could help improve the quality of life of couples affected by breast cancer.

ELIGIBILITY:
Inclusion Criteria:

-Patient has received a diagnosis within the last 5 years of invasive breast carcinoma (non- metastatic), or ductal carcinoma in-situ

* Patient has received a mastectomy or lumpectomy and undergone adjuvant therapy (i.e.

chemotherapy, radiation, tamoxifen)

* Patient is at least 1 month post-treatment.
* Couples are in a committed relationship of at least 3 months duration at the time of diagnosis
* Participants must be fluent in English
* Participants must be 80 years of age or younger
* Participants will require convenient access to a computer with a reliable internet connection in a private setting and have access to videoconferencing software (available for download at no cost).

Exclusion Criteria:

* One or both of the partners are currently struggling with any mental illness that would interfere with the ability to participate (e.g. actively suicidal; currently psychotic
* Couples who plan to participate in couples or sex counselling during the study
* Couples experiencing significant levels of relationship distress (e.g. presence of violence or abuse), in which case they will be referred for couple counseling

Max Age: 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Change in Sexual Function Questionnaire for Men and Women (SFQ-W, SFW-M) scores from pre (0 weeks) to post-treatment (6 weeks), and 3 month follow-up | pre-treatment (0 weeks), immediate post-treatment (6 weeks), and 3 month follow-up
  The SFQ assesses couples' sexual satisfaction and functioning. The SFQ will be used to assess change in couples' level of sexual functioning.

SECONDARY OUTCOMES:
Revised Dyadic Adjustment Scale (RDAS) | pre-treatment (0 weeks), immediate post-treatment (6 weeks), and 3 month follow-up
  The RDAS assesses couple's level of relationship satisfaction.
Maudsley Marital Questionnaire (marital sub-scale only) | pre-treatment (0 weeks), immediate post-treatment (6 weeks), and 3 month follow-up
  The Maudsley Marital Questionnaire assesses martial quality and happiness.
Profile of Mood States Short Form (POMS-SF) | pre-treatment (0 weeks), immediate post-treatment (6 weeks), and three months follow-up
  The POMS-SF assesses overall psychological adjustment.
Centre for Epidemiological Studies Depression Scale | pre-treatment (0 weeks), immediate post-treatment (6 weeks), and three months follow-up
  This measure assesses psychological adjustment, specifically with respect to depressive symptoms.
Generalized Anxiety Disorder Assessment (GAD-7) | pre-treatment (0 weeks), immediate post-treatment (6 weeks), and three months follow-up
  This measure assesses psychological adjustment, specifically with respect to anxiety
Breast Cancer Prevention Trial Symptom Checklist | pre-treatment (0 weeks), immediate post-treatment (6 weeks), and three months follow-up
  The BCPT measures commonly reported physical and psychological symptoms associated with breast cancer and associated treatments.
Spousal Skills Checklist | pre-treatment (0 weeks), immediate post-treatment (6 weeks), and three months follow-up
  The SSC measures partners' perceived support of their female partners

OTHER OUTCOMES:
Program Expectancy Questionnaire | Pre-treatment (0 weeks)
  The Program Expectancy Questionnaire will assess participants' expectations for the intervention, including the degree to which they believe the intervention will be effective.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Fergus, PhD, Principal Investigator — Toronto Sunnybrook Regional Cancer Centre
Locations (1):
- Sunnbrook Odette Cancer Centre, Toronto, Ontario, Canada